CLINICAL TRIAL: NCT06955299
Title: Changed Serum Levels of Sirtuin1 and Sirtuin3 and Their Correlations With Sleep Quality and Cognitive Function in the Patients With Chronic Insomnia Disorder
Acronym: SIRT1 SIRT3
Status: Completed | Type: Observational
Sponsor: Chaohu Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, GaoXia Liu, Master Degree Candidate, Chaohu Hospital of Anhui Medical University
Other Study IDs: 81671316
Record Dates: First submitted 2025-04-14; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-01

CONDITIONS: Chronic Insomnia Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to explore whether mitochondrial dysfunction exists in patients with chronic insomnia disorder. The main questions it aims to answer are :

* Do serum mitochondrial markers change in patients with chronic insomnia?
* Is there a relationship between serum mitochondrial markers and sleep and cognition in patients with chronic insomnia disorder? The researchers will compare serum mitochondrial marker levels among participants in the chronic insomnia group with those in the healthy group, and analyze the relationship between the markers and sleep and cognition of the participants.

Participants will:

* Complete polysomnography, the Pittsburgh Sleep Quality Index (PSQI), the Chinese-BeiJing version of the Montreal cognitive assessment (MoCA-C), the Blue Velvet Arena Test (BVAT), the Nine Box Maze Test (NBMT) to assess sleep and cognition.
* The venous blood was drawn to detect mitochondrial marker levels.

ELIGIBILITY:
Inclusion Criteria:

* meet the diagnostic criteria of the third edition of the International Classification of Sleep Disorders,26 At the same time, meet the following requirements: ① Duration suffered form insomnia > 6 months; ② 18-60 years old; ③ Receiving education ≥ 9 years of, without any understanding and hearing impairment; ④ The Pittsburgh Sleep Quality Index (PSQI) > 7 sores, Hamilton Anxiety Scale-14 (HAMA-14) < 14 scores, The Patient Health Questionnaire-9 (PHQ-9) < 10 scores; ⑤ There was no history of any sedative and hypnotic drugs in the two weeks prior to the visit

Exclusion Criteria:

* patients during pregnancy or breastfeeding or patients who have taken sedative hypnotic drugs or any other drugs that may affect sleep, mood and cognitive function within two weeks were not eligible for the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Qualified and voluntary subjects were recruited from the Sleep Disorder Department of Chaohu Hospital affiliated to Anhui Medical University from October 2021 to July 2023.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
The biological contents of SIRT1 and SIRT3 in all serum specimens were detected by enzyme-linked immunosorbent assay (ELISA) | Participants completed the assessment and PSG on the first day, and venous blood samples were collected at around 8 am on the next day for SIRT1 and SIRT3 detection
  All the test data were analyzed by SPSS26.0 statistical software, When P≤ 0.05 was considered statistically significant, two-sided test was conducted. Compared with the healthy group, the levels of SIRT1 (Z= -6.718,P<0.001) and SIRT3 (Z=-6.223,P<0.001) in the CID group were significantly increased.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Chaohu Hospital of Anhui Medical University, Hefei, Anhui, China